CLINICAL TRIAL: NCT03854747
Title: Investigation of the Effect of Cervical Spinal Stabilization Exercises on Spinal Posture, Cervical Proprioception and Postural Instability in Patients With Parkinson's Disease
Brief Title: The Effect of Cervical Spinal Stabilization Exercises in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: BElibol (Unknown); NKöse (Unknown); GYÇakmaklı (Unknown); SAksoy (Unknown); RGöçmen (Unknown)
Responsible Party: Principal Investigator, Emine Nur Demircan, Phsiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parkinson's disease treatment
Record Dates: First submitted 2019-02-16; First posted 2019-02-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- working group (Experimental)
  Interventions: Other: cervical spinal stabilization exercise

INTERVENTIONS:
Other: cervical spinal stabilization exercise — The cervical region is one of the most affected regions of the musculoskeletal system due to the intensive proprioceptors. Studies have shown that many position sense proprioceptors are over the deep group cervical muscles such as longus colitis and longus capitis. The deep group cervical muscles, which perform a dynamic ligament function, have an important role in maintaining the stability of the spine as well as the proprioceptive sense. In particular, proprioceptive receptors, which are commonly found in the deep suboccipital muscles; There are cervical and reflex connections with vestibular, visual and postural control systems.
  Arms: working group

SUMMARY:
Parkinson's disease (PH); it occurs due to dopamine deficiency due to the loss of dopaminergic neurons in a degenerative process in the substantia nigra found in the middle brain; resting tremor, bradykinesia, trunk and extremities rigidity, mask facial and postural instability characterized by a neurodegenerative disease. These findings are basic and also motor symptoms of Parkinson's Disease. Non-motor symptoms include many problems ranging from autonomic dysfunction to sensory symptoms.

Treatment of Parkinson's disease requires a multidisciplinary approach such as medical treatment, physiotherapy and rehabilitation, surgical treatment.

Physiotherapy programs applied to patients with Parkinson's disease include classical physiotherapy methods and neurophysiological based methods.

Spinal stabilization is an important concept for proper control of body balance and extremity movements. Spinal stabilization training was based on biomechanics, neurophysiology and physiotherapy research. Stabilization exercises, which form the basis of spinal stabilization training, increase the strength and endurance of the postural and stabilizing muscles using the basic principles of motor learning and improve stability control in stable and unstable positions, provides postural smoothness.

The cervical region is one of the most affected regions of the musculoskeletal system due to the intensive proprioceptors.

Although studies have been carried out to investigate the effect of spinal stabilization exercises in Parkinson's patients, there is no study on the effect of cervical region stabilization exercises in the literature despite these important connections of the cervical region.

For these reasons, this study is planned to investigate the effects of cervical spinal stabilization exercises on spinal posture, cervical proprioception and postural instability in Parkinson's patients.

Hypothesis 1: When cervical spinal stabilization exercises are added to the traditional physiotherapy program in Parkinson's patients, it will be more effective in correcting spinal posture.

Hypothesis 2: When cervical spinal stabilization exercises are added to the traditional physiotherapy program in Parkinson's patients, cervical proprioception will develop better.

Hypothesis 3: In the case of Parkinson's patients, when the cervical spinal stabilization exercises are added to the traditional physiotherapy program, postural stability may be more pronounced.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease,
* Having planned a traditional physiotherapy program for Parkinson's disease and referring to Hacettepe University Faculty of Health Sciences Physiotherapy and Rehabilitation Department,
* 40 to 80 years old,
* According to Hoehn-Yahr scale to be in stage 2 or 3,
* Having scored 30 points above the posture evaluation
* Postural disorder in the femoral region, but the absence of structural disorder (congenital spinal deformities in medical evaluations prior to the study, structural disorders caused by other diseases should be determined that the spine does not have problems),
* 26 points higher than the mini-mental test,
* Disease duration is 3 years and above,
* The absence of any other neurological disease other than vestibular and / or Parkinson's, which may affect muscle strength, balance and coordination,
* Spinal colon and lower extremity musculoskeletal system, which may affect the stabilization of any surgery has been identified as.

Exclusion Criteria:

* Volunteers who do not comply with the inclusion criteria will not be included in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Static Posturography | baseline to 8 week after
  balance measurement (Number of Participants estimated 20 individuals)
X-Ray Measure | baseline to 8 week after
  scoliosis graphy
Bubble Inclinometer | baseline to 8 week after
  measurement of spine curvature angle (Number of Participants estimated 20 individuals)
Scoliometer | baseline to 8 week after
  measurement of spine curvature angle
UPDRS | baseline to 8 week after
  Unified Parkinson's Disease Rating Scale. There are 4 sub-parameters. 1. mental status, behavior and mental state 2. daily life activities 3. motor inspection 4. treatment complications. mental status, behavior and mental state total 16 points, daily activity total 52 points, Motor parameter total 92 points, treatment complications total 23 points. Total maximum 183 points. the total score is calculated by adding all sub-parameter scores. low value is good, high value is a symptom of bad result.
Berg Balance Scale | baseline to 8 week after
  balance measurement. It is a 14-item balance scale. The range of points is between 0 and 56. The total score is calculated by summing the points of each item. high score good balance, low score indicates bad balance.
Posture Analyse | baseline to 8 week after
  is a scale that evaluates the participant's 13 different regions from posterior and lateral to postural disorder. the scoring of each region is 1-3-5. if normal is 5 points, moderate level is 3 points, if there is any advanced disorder 1 point is given. the total score is determined by summing all the values. total maximum 65, minimum 13 points. high score good posture, low score indicates bad posture
Cervical Proprioception | baseline to 8 week after
  A tool used to evaluate the sense of proprioception in the cervical region of the participants with the Cervical Range of Measure(CROM) device
Visual Analog Scale | baseline to 8 week after
  Visual Analog Scala. Numerical rating scale of pain intensity. 0 to 10 is a scale with a rating. 0 points no pain 10 points is a scale with very severe pain. the participant is asked to say a value in this range according to the severity of pain.
10 meter walk test | baseline to 8 week after
  walking speed calculation
Timed Get up and Walk Test | baseline to 8 week after
  walking time and cadence calculation
Cervical Ventral Endurance Evaluation | baseline to 8 week after
  Endurance evaluation will be done to deep cervical flexor extensor muscles
Muscle Strength Assessment | baseline to 8 week after
  evaluation of the strength of the muscles in the cervical region and shoulder circumference
Evaluation of Muscle Shortness | baseline to 8 week after
  measurement of shortness of some muscles in upper extremity and lower extremity with goniometer and tape measure
Normal Joint Movement Assessment | baseline to 8 week after
  measurement of normal range of motion
Short Form-36 | baseline to 8 week after
  SF-36 (Short Form 36). Quality of life survey. examines 8 dimensions of health with 36 items. physical function, social function, role restrictions, mental health, vitality, pain and general health. The scores of each parameter are between 0 and 100. 0 bad, 100 good results. is calculated by taking the values of the sub-parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kay TM, Gross A, Goldsmith CH, Rutherford S, Voth S, Hoving JL, Bronfort G, Santaguida PL. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD004250. doi: 10.1002/14651858.CD004250.pub4. PMID 22895940
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Park A, Stacy M. Non-motor symptoms in Parkinson's disease. J Neurol. 2009 Aug;256 Suppl 3:293-8. doi: 10.1007/s00415-009-5240-1. PMID 19711119
- [Background] Shujaat F, Soomro N, Khan M. The effectiveness of Kayaking exercises as compared to general mobility exercises in reducing axial rigidity and improve bed mobility in early to mid stage of Parkinson's disease. Pak J Med Sci. 2014 Sep;30(5):1094-8. doi: 10.12669/pjms.305.5231. PMID 25225533
- [Background] Carter JM, Beam WC, McMahan SG, Barr ML, Brown LE. The effects of stability ball training on spinal stability in sedentary individuals. J Strength Cond Res. 2006 May;20(2):429-35. doi: 10.1519/R-18125.1. PMID 16686575
- [Background] Kaya DO, Ergun N, Hayran M. Effects of different segmental spinal stabilization exercise protocols on postural stability in asymptomatic subjects: randomized controlled trial. J Back Musculoskelet Rehabil. 2012;25(2):109-16. doi: 10.3233/BMR-2012-0318. PMID 22684202
- [Derived] Demircan EN, Kose N, Cakmakli GY, Aksoy S, Gocmen R, Zengin HY, Elibol B. Do cervical stabilization exercises change the effects of conventional exercises in patients with Parkinson's disease? Neurol Res. 2023 Oct;45(10):936-946. doi: 10.1080/01616412.2023.2249699. Epub 2023 Aug 22. PMID 37608568